CLINICAL TRIAL: NCT02012673
Title: The Safety and Feasibility of Re-treating Patients With Severe Emphysema With the RePneu LVRC System: a Pilot Study.
Brief Title: A Safety and Feasibility Study of Re-treating Patients With Severe Emphysema With the RePneu LVRC System.
Acronym: RECOIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, MD PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECOIL-study
Record Dates: First submitted 2013-09-04; First posted 2013-12-16 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: COPD; Emphysema
Keywords: COPD; Emphysema; Bronchoscopy; Lung Volume Reduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bronchoscopic lung volume reduction (Experimental): Bronchoscopic lung volume reduction with the RePneu Lung Volume Reduction Coil system
  Interventions: Device: Bronchoscopic lung volume reduction

INTERVENTIONS:
Device: Bronchoscopic lung volume reduction — Bronchoscopic lung volume reduction with the RePneu Lung Volume Reduction Coil system. The RePneu LVRC is an implantable device, delivered through a fiber-optic bronchoscope, designed specifically to treat patients suffering from emphysema. The Coil is intended to compress the most damaged parenchyma and tension the surrounding tissue, which increases elastic recoil, reduces hyperinflation and redirects air to healthier portions of the lung for more effective ventilation.

SUMMARY:
Rationale:

The combined data from 3 studies outside the Unites States investigating the Lung Volume Reduction Coil system (RePneu LVRC) showed statistically significant improvements in pulmonary function, exercise capacity and quality of life at both 6-Months and 12-Months post treatment. 24 months post treatment the improved pulmonary function and exercise capacity are slightly decreasing. Retreating the patient with the LVR coil system in other parts of the lung could potentially lead to new improvements in lung function, dyspnea, exercise capacity and quality of life and may reduce the rate of decline.

Objective:

To investigate the safety and feasibility of re-treating patients with severe Chronic Obstructive Pulmonary Disease (COPD) with the RePneu LVRC system.

DETAILED DESCRIPTION:
Rationale:

The combined data from 3 studies outside the Unites States investigating the Lung Volume Reduction Coil system (RePneu LVRC) showed statistically significant improvements in pulmonary function, exercise capacity and quality of life at both 6-Months and 12-Months post treatment. 24 months post treatment the improved pulmonary function and exercise capacity are slightly decreasing. Retreating the patient with the LVR coil system in other parts of the lung could potentially lead to new improvements in lung function, dyspnea, exercise capacity and quality of life and may reduce the rate of decline.

Objective:

To investigate the safety and feasibility of re-treating patients with severe Chronic Obstructive Pulmonary Disease (COPD) with the RePneu LVRC system.

Study design:

This study is a non randomized uncontrolled intervention.

Study population: Patients with severe emphysema who have previously been treated with the lung volume reduction coil system and significantly improved in lung function, exercise capacity or quality of life, 6 months after the treatment.

Intervention:

Patients will receive a lung volume reduction coil treatment by bronchoscopy.

Main study parameter:

The safety objective of this study is to identify the potential number and type of device-related and procedure-related adverse effects.

Secondary study parameters:

Lung function

* Change in RV, 6 months following treatment
* Change in RV/TLC ratio, 6 months following treatment
* Changes in FEV1 and FVC, 2 and 6 months following treatment

Quality of life

* Change in the SGRQ score, 2 and 6 months following treatment
* Change in the CCQ score, 2 and 6 months following treatment

Functional measures

* Change in the mMRC score, 2 and 6 months following treatment
* Change in the 6MWD, 2 and 6 months following treatment

ELIGIBILITY:
Inclusion Criteria:

1. Treated with the RePneu LVRC system > 24 months ago.
2. Six months after the first bilateral treatment with the RePneu LVRC system the patient had a significant improvement above the established minimal important difference (MID) of 6-minute walk distance (6MWD: 26 meter) or of forced expiratory volume in 1 second (FEV1: 100ml) or of St. Georges Respiratory Questionnaire total score (SGRQ: 4 points).
3. Subject has marked dyspnea scoring ≥2 on mMRC scale of 0-4.
4. Subject has stopped smoking for at least 6 months prior to entering the study.
5. Subject read, understood and signed the Informed Consent form.
6. Subject has completed a pulmonary rehabilitation program within 6 months prior to treatment and/or regularly performing maintenance respiratory rehabilitation if initial supervised therapy occurred more than 6 months prior to baseline testing.
7. Subject has received Influenza vaccinations consistent with local recommendations and/or policy.

Exclusion Criteria:

1. Subject has co-morbidities that may significantly reduce subject's ability to improve exercise capacity (e.g., severe arthritis, planned knee surgery) or baseline limitation on 6MWT is not due to dyspnea.
2. Subject has severe gas exchange abnormalities as defined by:

   PaCO2 >8.0 kPa; PaO2 < 6.0 kPa (room air).
3. Subject has a history of recurrent clinically significant respiratory infections, defined as 3 hospitalizations for respiratory infection during the year prior to enrollment.
4. Subject has severe pulmonary hypertension defined by right ventricular systolic pressure >50 mm Hg via echocardiogram.
5. Subject has an inability to walk >140 meters in 6 minutes.
6. Subject has evidence of other severe disease (such as, but not limited to, lung cancer or renal failure), which in the judgment of the investigator may compromise survival of the subject for the duration of the study.
7. Subject is pregnant or lactating, or plans to become pregnant within the study timeframe.
8. Subject has an inability to tolerate bronchoscopy under moderate sedation or general anesthesia.
9. Subject has clinically significant bronchiectasis.
10. Subject has giant bullae >1/3 lung volume.
11. Subject has had previous LVR surgery, lung transplantation or lobectomy.
12. Subject has been involved in pulmonary drug or device studies within 30 days prior to this study.
13. Subject is taking >20 mg prednisone (or equivalent dose of a similar steroid) daily.
14. Subject requires high level chronic immunomodulatory therapy to treat a moderate to severe chronic inflammatory autoimmune disorder.
15. Subject is on an antiplatelet (such as Plavix) or anticoagulant therapy (such as heparin or Coumadin) which cannot be stopped for 7 days prior to procedure.
16. Subject has a sensitivity or allergy to Nickel.
17. Subject has a known sensitivity to drugs required to perform bronchoscopy.
18. Subject has any other disease, condition(s) or habit(s) that would interfere with completion of study and follow up assessments, would increase risks of bronchoscopy or assessments, or in the judgment of the investigator would potentially interfere.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number and type of adverse effects as a measure of safety between baseline and 6 months follow up | Baseline - 6 month follow up
  The safety objective of this study is to identify the potential number and type of device-related and procedure-related adverse effects.

SECONDARY OUTCOMES:
Change from Baseline in Lung function at 2 months | Baseline vs 2 month follow up
  -Changes in FEV1 and FVC, 2 months following treatment
Change from Baseline in Quality of life at 2 months | Baseline vs 2 month follow up
  * Change in the SGRQ score, 2 months following treatment
  * Change in the CCQ score, 2 months following treatment
Change from Baseline in functional measures at 2 months | Baseline vs 2 month follow up
  * Change in the mMRC score, 2 months following treatment
  * Change in the 6MWD, 2 months following treatment
Change from Baseline in Lung function at 6 months | Baseline vs 6 month follow up
  * Change in RV, 6 months following treatment
  * Change in RV/TLC ratio, 6 months following treatment
  * Changes in FEV1 and FVC, 6 months following treatment
Change from Baseline in quality of life at 6 months | Baseline vs 6 month follow up
  * Change in the SGRQ score, 6 months following treatment
  * Change in the CCQ score, 6 months following treatment
Change from Baseline in functional measures at 6 months | Baseline vs 6 month follow up
  * Change in the mMRC score, 6 months following treatment
  * Change in the 6MWD, 6 months following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — University Medical Center Groningen, Department of Pulmonary Diseases
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands